CLINICAL TRIAL: NCT06790394
Title: A Test-retest Study to Evaluate the Reproducibility of [18F]Florbetaben PET Imaging in Patients With Cardiac Amyloidosis and Control Patients
Brief Title: Test-retest Study With [18F]FBB in Cardiac Amyloidosis
Acronym: CATI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging GmbH (Industry)
Collaborators: pharmtrace (Unknown)
Responsible Party: Sponsor
Organization: Life Molecular Imaging SA (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FBB-02-01-24
Record Dates: First submitted 2024-12-19; First posted 2025-01-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with cardiac disease (Experimental): All eligible AL, ATTR and non-CA patients will receive two injections of the investigational imaging agent florbetaben: at a baseline PET imaging session and at a follow-up PET imaging session to evaluate the test-retest imaging characteristics. 5 patients of each group will be required.
  Interventions: Drug: Florbetaben F18

INTERVENTIONS:
Drug: Florbetaben F18 — Florbetaben F18 is a radioactive diagnostic agent being developed for the indication of PET imaging of the heart to detect amyloid pathology. All patients will receive two administrations of Florbetaben F18 at a radioactive dose of 300 megabecquerel (MBq).

SUMMARY:
This study is an open-label study to evaluate and characterize test-retest reliability of [18F]florbetaben PET in subjects with AL-CA and ATTR-CA compared to non-CA subjects. Quantification of the [18F]florbetaben parameters related to the deposition of amyloid in the heart (such as Myocardial Tracer Retention (MTR) or Retention Index (RI)), and the variability in these parameters after repeated imaging will be evaluated. Measurement of blood metabolites and comparison of invasive with non-invasive quantification of [18F]florbetaben uptake in the heart will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria (for all subjects):

  * Males and females aged ≥40 years
  * Able to understand, sign, and date written informed consent
  * Written informed consent must be obtained before any assessment is performed
  * Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or post-menopausal for at least 1 year (no menses for 12 months without an alternative medical cause). If they are of child-bearing potential, they must commit to use of a highly effective contraceptive measure for one week after the PET scan (including combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence)
  * Male subjects and their partners of childbearing potential must commit to the use of a highly effective method of contraception for a minimum of 90 days following each PET scan (including, for female partners of childbearing potential, combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, male subjects with vasectomy or sexual abstinence)
  * Male subjects must commit to not donate sperm for a minimum of 90 days after the PET scan
  * Medications taken for treatment of multiple myeloma or chronic diseases of the heart or tafamides treatment are maintained on a stable dosage regimen.
  * Patients on stable coagulation, if arterial blood sampling isperformed.
* Inclusion criteria for AL-CA and ATTR-CA patients:

  • Patients with a clinical diagnosis of cardiac AL amyloidosis or cardiac ATTR diagnosis according to diagnostic criteria
* Inclusion criteria for control patients:

The control subjects must meet one of the following criteria:

* Patients without heart failure and no suspicion of cardiac amyloidosis OR
* Patients with impaired heart function but cardiac amyloidosis ruled out by echocardiography, CMR or cardiac biopsy OR
* Patients with known plasma cell dyscrasia (MGUS, multiple myeloma) but no clinical signs of cardiac amyloidosis detected by echocardiography or CMR

Exclusion Criteria:

* Subject has received, in the last 3 months, or currently receives amyloid targeting monoclonal antibody therapy.
* Any known allergic reactions or hypersensitivity towards any compound of the study drug
* Hemoglobin value < 10 g/dL
* Severe hepatic impairment (AST or ALT >5 x ULN; bilirubin >3 x ULN)
* Subject receives hemodialysis or peritoneal dialysis
* Inability to lay flat for up to 60 min
* Pregnant, lactating or breastfeeding
* Unwilling and/or unable to cooperate with study procedures
* Having received a PET scan within one week before the 18F]florbetaben PET scan
* For patients were arterial sampling isperformed: Subject has a contraindication to arterial cannulation, including but not limited to allergy to local anesthetics, peripheral vascular disease, Raynaud's phenomenon as determined by abnormal Allen's test or abnormal coagulation profile at screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Test-Retest variability of cardiac [18F]florbetaben PET uptake | The duration of the study for participants may be up to 73 days.
  Percent Test-Retest variability (%) of cardiac 18F florbetaben PET

SECONDARY OUTCOMES:
Test-Retest variability of extracardiac [18F]florbetaben uptake | The duration of the study for participants may be up to 73 days.
  Percent Test-Retest variability (%) of extracardiac 18F forbetaben PET
Net influx rate derived from full tracer kinetic modelling | The duration of the study for participants may be up to 73 days.
  Net influx rate Ki [ml/cm3/min]
Volume of distribution derived from full tracer kinetic modelling | The duration of the study for participants may be up to 73 days.
  Volume of distribution Vd
Safety and tolerability of [18F]florbetaben | The duration of the study for participants may be up to 73 days.
  Number of participants with treatment-related adverse events as assessed by CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Free Hospital, London
  - King's College London, London